CLINICAL TRIAL: NCT03302728
Title: A Phase 1b Study of Brentuximab Vedotin and Lenalidomide in Patients With Relapsed/ Refractory Cutaneous T-cell Lymphoma, CD30-positive Peripheral T-cell Lymphoma, or CD30-positive Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Lenalidomide in Patients With Relapsed/ Refractory T-cell Lymphoma or Hodgkin Lymphoma
Acronym: EpiBrentlen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/34
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Hodgkin Lymphoma
Keywords: CD 30 positive, relapsed, refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell, Peripheral; Hodgkin Disease; Recurrence | interventions — Lenalidomide; Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: This is a single arm dose escalation study. There are four dose levels for the combination of Brentuximab vedotin and Lenalidomide considered during the dose escalation.
  Starting Dose Level 1: Brentuximab vedotin 1.8mg/kg q21 days & Lenalidomide 15 mg daily (D1-14)
  The dose can be decreased as follows:
  Level -2 Brentuximab vedotin 1.2mg/kg q21 days & Lenalidomide 5 mg daily (D1-14)
  Level -1 Brentuximab vedotin 1.2mg/kg q21 days & Lenalidomide 10 mg daily (D1-14)
  or the dose can be escalated as follows:
  Level 2 Brentuximab vedotin 1.8mg/kg q21 days & Lenalidomide 25 mg daily (D1-14)
  Patients will be assigned a starting dose by the safety committee; this will be communicated by the PI and/or their designated sub-investigator prior to planned Cycle1 Day 1 for each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenalidomide & brentuximab vedotin (Experimental): Brentuximab vedotin 1.8mg/Kg Lenalidomide 15 mg
  Interventions: Drug: Lenalidomide 15mg; Drug: Brentuximab Vedotin 1.8 mg/Kg

INTERVENTIONS:
Drug: Lenalidomide 15mg — At commencement of study : Lenalidomide will commence at 15 mg daily for days 1-14 of each cycle. Maximum number of cycles = 16. This is a dose finding study so doses will be adjusted depending on toxicity assessment over the course of the study. Dose may vary from 5 mg -25 mg daily depending on dose escalation results and recommendation of safety committee
  Other Names: Revlimid
Drug: Brentuximab Vedotin 1.8 mg/Kg — At commencement of study : Brentuximab vedotin 1.8mg/kg IV on day 1, repeated every 21 days. Maximum number of cycles = 16. This is a dose finding study so doses will be adjusted depending on toxicity assessment over the course of the study. Dose may be either 1.2 mg/Kg q21 days or 1.8 mg/kg q21 days depending on dose escalation results and recommendation of safety committee
  Other Names: Adcetris

SUMMARY:
This study is investigating the combination of Brentuximab vedotin and lenalidomide in the treatment of relapsed/refractory peripheral T cell lymphoma or cutaneous T cell lymphoma or Hodgkin lymphoma.

It is hypothesised that lenalidomide may augment the actions of Brentuximab vedotin in these patient groups. The primary objective of the study is to determine the maximum tolerated dose of the combination treatment, which can be used in subsequent studies. The study will also investigate disease response and survival.

Participants will receive Brentuximab vedotin (once every 21 days i.e. 1 cycle) and lenalidomide (daily from day 1 -14 of each cycle) for a maximum of 48 weeks and will be followed for a subsequent 6 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18 years or older.
2. Patient must have a diagnosis of a CD30+ Hodgkin Lymphoma or CD30+ peripheral T-cell lymphoma. Patients with either Hodgkin lymphoma or T-cell lymphoma must have expression of CD30 in ≥10% of lymphoma cells. Patients with CTCL will be considered for inclusion even if CD30 immunohistochemical staining with BerH2 antibody is low or negligible (<10%).

   1. Peripheral T-cell lymphoma: patients must be considered relapsed or refractory after at least one prior chemotherapeutic regimen or be considered by the investigator to be not suitable for chemotherapy
   2. Cutaneous T-cell lymphoma: patients must be relapsed or refractory to one prior systemic therapy or be considered by the investigator to be not suitable for chemotherapy
   3. Patients with Hodgkin lymphoma and one of the following:

   i. Relapsed or refractory after at least 2 prior chemotherapy-containing regimens ii.Considered unsuitable for chemotherapy
3. Voluntary written informed consent must be given before performance of any study- related procedure.
4. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
5. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
6. Performance status of ECOG ≤2.
7. Clinical laboratory values as specified below. Blood tests must be within 10 days of patient registration:

   * Absolute neutrophil count >1.5 x109/L, or >1.0 x109/L in the setting of known marrow involvement by tumour.
   * Platelet count ≥75x109/L.
   * Total bilirubin must be < 1.5 x the upper limit of the normal (ULN) unless the elevation is known to be due to Gilbert syndrome.
   * ALT or AST must be < 2.5 x the upper limit of the normal range. AST or ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of haematologic/solid tumor in liver.
   * Serum creatinine must be < 150 µmol/L and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute.
   * Haemoglobin must be ≥ 80g/L.
8. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy (except alopecia) prior to registration.

Exclusion Criteria:

1. Female patients who are both lactating and breast-feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on planned cycle 1, day 1 prior to first dose of study drug.
2. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol.
3. Symptomatic neurologic disease compromising normal activities of daily living or requiring medication/s, including signs or symptoms of Progressive Multifocal Leucoencephalopathy (PML).
4. Any sensory or motor peripheral neuropathy greater than or equal to Grade 2 at registration.
5. Known history of any of the following cardiovascular conditions

   1. New York Heart Association (NYHA) Class III or IV heart failure (see Appendix 18.1).
   2. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
   3. A left-ventricular ejection fraction <50%
6. Any active systemic viral, bacterial, or fungal infection requiring systemic intravenous antibiotics or systemic antifungal therapies within 2 weeks prior to registration.
7. Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment.
8. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin or lenalidomide.
9. Known human immunodeficiency virus (HIV) positive.
10. Known hepatitis B surface antigen (HBsAg)-positive, or known or suspected active hepatitis C infection. Patients who are Hepatitis B core antibody positive with no evidence of active disease, i.e.

    HBsAg negative/ negative hepatitis B viral load, will still be considered eligible for inclusion, but must receive viral suppressive therapy for the duration of the trial.
11. Active systemic malignancy likely to require treatment within the next two years, or previous diagnosis of another malignancy with residual disease. Patients with non-melanoma skin cancer or carcinoma- in-situ of any type are not excluded if they have undergone complete resection.
12. Previous exposure to brentuximab vedotin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended phase 2 dose (RP2D) of the combination of lenalidomide and brentuximab vedotin | 70 weeks
  Maximum tolerated dose, dose-limiting toxicities of the combination therapy, and recommended phase 2 dose, in patients with relapsed/refractory cutaneous T-cell lymphoma, CD30-positive Hodgkin lymphoma and CD30-positive peripheral T-cell lymphoma. The MTD is defined as the highest dose level at which the incidence of DLT was less than 33%.

SECONDARY OUTCOMES:
Safety profile of the combination of lenalidomide and brentuximab vedotin | 70 weeks
  Toxicities measured using CTCAE V4.03.
Treatment intensity. | 48 weeks
  Treatment intensity defined as the actual total dose received divided by the actual treatment period.
Objective response rate | 70 weeks
  Objective response, defined as achieving either complete response (CR) or partial response (PR) at some stage from time of commencement of treatment until conclusion of period of follow-up (maximum 16 cycles of treatment followed by 6 months of follow-up), or until time of documented progressive disease (defined as clinical and/or radiologic progression).
Cytostatic response. | 70 weeks
  Cytostatic response, defined as achieving complete response (CR), partial response (PR) or stable disease (SD) lasting >6 months from time of commencement of treatment until progressive disease (PD).
Event free survival. | 70 weeks
  Event free survival (EFS), defined as the time from commencement of treatment to date of early discontinuation of treatment due to toxicity, date of documented disease progression at any site, or date of death from any cause, whichever occurs first.
Overall survival | 70 weeks
  Overall survival (OS), defined as the time from commencement of treatment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Dr, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No